CLINICAL TRIAL: NCT05218356
Title: Phase IIa Randomized Placebo Controlled Clinical Study of Codivir in Hospitalized Patients with Moderate COVID-19
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Code Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-21-01
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Electrocardiography; Restraint, Physical

STUDY DESIGN:
Intervention Model Description: This is a double-blind, multicentre, multinational study to evaluate the safety and collect preliminary efficacy data of Codivir drug product in 130 hospitalized adults with moderate COVID-19 symptoms. COVID-19 symptoms (fever, cough, myalgia and changes in smell or taste) onset must be within 7 days prior enrolment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the study is a double-blind study: neither the participants nor the investigators will be aware of arm allocation of each study participant. Blindness is important to avoid bias. Monitoring and reporting of the success of blindness are important for the reader's confidence of the trial results. Groups should be marked by capital letter and blindness should maintain throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Codivir treatment (Experimental): 20 mg administrated by subcutaneous (SC) injection, twice a day, for 7 days
  Interventions: Drug: Covidir injections; Diagnostic Test: Quantitative PCR SARS-CoV-2; Diagnostic Test: IgM and IgG dosage; Diagnostic Test: Screening Blood tests; Diagnostic Test: Electrocardiogram; Other: NEWS-2 score; Other: WHO score; Other: Physical examination; Other: COVID-19-Related Symptoms assessment
- Placebo treatment (Placebo Comparator): Placebo administrated in subcutaneous (SC) injection, twice a day, for 7 days
  Interventions: Drug: Covidir injections; Diagnostic Test: Quantitative PCR SARS-CoV-2; Diagnostic Test: IgM and IgG dosage; Diagnostic Test: Screening Blood tests; Diagnostic Test: Electrocardiogram; Other: NEWS-2 score; Other: WHO score; Other: Physical examination; Other: COVID-19-Related Symptoms assessment

INTERVENTIONS:
Drug: Covidir injections — administration of the investigational product CODIVIR/Placebo at a dose of 20 mg twice a day subcutaneously at visits Day0-Day6 (7 days total)
  Other Names: Experimental drug administration
Diagnostic Test: Quantitative PCR SARS-CoV-2 — detection of viral RNA in nasopharyngeal and oropharyngeal samples by the Real Time Protein Chain Reaction technique.
Diagnostic Test: IgM and IgG dosage — lood collection for dosage of Anti SARS-CoV-2 antibodies.
Diagnostic Test: Screening Blood tests — omplete blood count, urea, creatinine, uric acid, sodium, potassium, chloride, calcium, glucose, glycated hemoglobin, alkaline phosphatase (FA), alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubins and fractions ( BTF), total proteins and fractions (PTF), lipid profile (total cholesterol, fractions and triglycerides); coagulogram (TP, aPTT); D-dimer; C-reactive protein; HIV, HBV, HCV serology; Ferritin; troponin, fibrinogen,Coagulogram (TP, aPTT); D-dimer, Pregnancy test for non-sterile women.
Diagnostic Test: Electrocardiogram — valuation by the principal investigator or assistant physician with a complete physical examination
  Other Names: ECG
Other: NEWS-2 score — assessment of the participant by the NEWS-2 score.
Other: WHO score — assessment of the participant by the score of the World Health Organization.
Other: Physical examination — evaluation by the principal investigator or assistant physician
Other: COVID-19-Related Symptoms assessment — will be completed by the study staff member based on patient status and answers.

SUMMARY:
This is a double-blind, multicentre, multinational study to evaluate the safety and collect preliminary efficacy data of Codivir drug product in 130 hospitalized adults with moderate COVID-19 symptoms. COVID-19 symptoms (fever, cough, myalgia and changes in smell or taste) onset must be within 7 days prior enrolment. Treatment will begin in the hospital, participants will be discharged according to medical decision and continue the treatment until to Day 7 at home and followed up to day 28.

DETAILED DESCRIPTION:
eligible hospitalized participants will be recruited to the study and will receive standard of care treatments as well as Codivir or placebo, which will be administered at a dose of 20 mg SC, twice a day, for 7 days. If up to medical decision of the medical staff in the site, the patient should be released before Day 7, site study team will contact the medical monitor of the study to get the instructions. Participants will be followed up to the 28th day via phone contact. The phone visit will be performed to monitor the clinical symptoms, collect adverse events and concomitant medication and provide the patient with additional instructions, if relevant.

If they have progressed well, they will continue the treatment up to Day 7 at home, receiving a nurse's home visit twice a day to administer Codivir and collect vital signs. Participants will be followed up to Day 28 by telemedicine. A doctor will call them periodically to monitor the clinical evolution, collect adverse events, concomitant medication and instruct the participants. In case of unfavorable evolution, the participants will remain hospitalized receiving the appropriate care. The investigator will decide whether or not the investigational medication will continue, considering the participant's health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Male or female
* SARS-CoV-2 infection indicated by confirmed RT-PCR test
* Moderate hospitalized COVID-19 (at least two out of three criterias below):

  * Evidence of lower respiratory disease during clinical assessment (cough, fever, difficulty breathing) or imaging (X-rays)
  * Oxygen saturation (SpO2) in room air < 93%
  * <30 breaths per minute
* No signs of hemodynamic decompensation
* Absence of pregnancy in women of childbearing age
* Ability to understand and comply with the requirements of the protocol
* Consent to participate
* Consent to use at least one highly effective contraception methods (condoms, IUD, oral contraceptives) since the ICF signature and at least 30 days after the study.

Exclusion Criteria:

* Patients receiving oxygen supplementation except of nasal prongs, nasal intermittent positive pressure ventilation (NIPPV) or high flow nasal cannula (HFNC) that are allowed to be enrolled to the study).
* Positive RT-PCR test more than 72 hours prior to enrolment.
* Onset of symptoms more than 7 days prior to enrolment.
* Participant using drugs that are under clinical investigation in last 30 days.
* Body mass index less than 19.9 or greater than 35.
* Comorbidities such as: other serious infections, active malignancies, autoimmune diseases, liver, kidney or heart failure; another systemic disease and / or laboratory abnormality, which, in the investigator's opinion, prevent the patient from participating in the study.
* Concomitant HIV, HBV or HCV infection.
* Pregnancy or lactation.
* Vaccination for any other infection in the 4 weeks prior to enrolment.
* Any condition that increases the risk of participating in the study, in the opinion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Change in World Health Organization Ordinal Scale for clinical improvement | up to 28 days
  change in World Health Organization Ordinal Scale for clinical improvement in the treatment group in comparison with Placebo. the scale min score - 0 and max score - 8. the higher the scores mean a worse outcome

SECONDARY OUTCOMES:
Change in COVID-19-Related Symptoms score (measured on days 7, 14, 21, 28) in the treatment group in comparison with Placebo). | up to 28 days
  Each symptom is scored individually using the following response options and scoring values: Items 1-10: None = 0; Mild = 1; Moderate = 2; and Severe = 3 Items 11 and 12: Not at all = 0; 1-2 times = 1; 3-4 times = 2; 5 or more times = 3 Items 13 and 14: Sense of smell/taste same as usual = 0; Sense of smell/taste less than usual = 1; No sense of smell/taste = 2. he higher the scores mean a worse outcome
adverse events | up to 28 days
  Incidence and severity of adverse events related to the investigational product in the treatment group in comparison with Placebo
RT-PCR viral load | up to 28 days
  Time to decreased RT-PCR viral load in the treatment group in comparison with Placebo
IgM & IgG anti-SARS-CoV-2 | up to 28 days
  Evolution of IgM & IgG anti-SARS-CoV-2 in the treatment group in comparison with Placebo

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Hospital de Amor, Paulo Prata, Barretos/SP/BRA
  - Infection Control, Prado, Belo Horizonte/MG/BRA
  - Instituto Lobus, Casa de Pedra, Volta Redonda/RJ/BRA
  - A2Z Clinical, Vila Martina, Volta Redonda/RJ/BRA
  - Casa de Saude, Centro

IPD SHARING:
Plan to Share IPD: No